CLINICAL TRIAL: NCT03028064
Title: Point of Care Testing of Platelet Function in Patients With Acute Upper Gastrointestinal Bleeding
Acronym: POCGIB
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Other Study IDs: POCGIB
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Hematemesis; Melena; Gastrointestinal Hemorrhage; Platelet Dysfunction
MeSH Terms: conditions — Hematemesis; Melena; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: blood taking — in this cohort study, we will take blood to examine the platelet function

SUMMARY:
Acute upper gastrointestinal bleeding (AUGIB) is a common medical emergency. In an ageing population, antiplatelet drugs are increasingly being prescribed for treatment and prophylaxis against cardiovascular thrombo-embolic events. In many patients, platelet dysfunction mostly acquired is the principal cause of bleeding. To clinicians, the management of patients on antiplatelet drugs or anticoagulants is a challenge. One has to carefully balance the bleeding against thrombo-embolic risks. Therefore measuring platelet function should be integral in the management plan. A quantitative measurement allows titration of platelet function in accordance with bleeding or thromboembolic risk. Platelet function has not been studied in a large cohort of patients with acute upper gastrointestinal bleeding. As a first step, the study will determine if platelet dysfunction is associated with clinical outcome. In this prospective, observational single centre cohort study of consecutive patients with overt signs of acute upper gastrointestinal bleeding, their platelet function by point of care tests (light transmittance aggregometry, verify now p2y12,the platelet function analysis system (PFA-100) upon their admissions. Patients will be followed up for 30 days after trial enrollment. The primary endpoint is defined as significant bleeding that requires interventions (endoscopic, radiologic or surgery). Secondary end points include cardio- and cerebrovascular thrombo-embolic events and all cause deaths. A receiver operating characteristic (ROC) curve analysis is calculated for each point-of-care test to evaluate if individual test can distinguish between patients with and without primary end point. This study aims to evaluate the capability of platelet function tests to predict clinical outcome in patients with AUGIB. Logistic regression models will then be built in search for independent correlates to the primary and secondary endpoints and to adjust for confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* patients with overt signs of acute upper gastrointestinal bleeding (melena, coffee ground or fresh hematemesis with or without circulatory instability)

Exclusion Criteria:

* asymptomatic patients with anemia are absence of positive gastroscopic findings to support gastrointestinal bleeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with overt signs of acute upper gastrointestinal bleeding (melena, coffee ground or fresh hematemesis with or without circulatory instability)
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Active bleeding that requires interventions (endoscopic, radiologic or surgery) | within 30 days of trial inclusion
  Data on whether patients experience further bleeding that requires interventions, the type of interventions and the time of further bleeding after trial inclusion, will be collected through electronic medical record

SECONDARY OUTCOMES:
All cause deaths, cardiovascular or cerebral thrombotic events | within 30 days of trial inclusion
  All cause deaths, cardiovascular or cerebral thrombotic events

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Centre, Hong Kong, HONG KONG, China

IPD SHARING:
Plan to Share IPD: Undecided